CLINICAL TRIAL: NCT05754073
Title: A Randomized, Double-blind, Placebo-controlled Study of Intranasal Oxytocin for Bone Health in Children With Autism Spectrum Disorder
Brief Title: Oxytocin Effects on Bone in Children With Autism Spectrum Disorder
Acronym: BOX
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Elizabeth Austen Lawson (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); University of Virginia (Other)
Responsible Party: Sponsor-Investigator, Elizabeth Austen Lawson, Director of the Interdisciplinary Oxytocin Research Program, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2023P000307
Record Dates: First submitted 2023-02-22; First posted 2023-03-03 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2024-12

CONDITIONS: Autism Spectrum Disorder; Bone Health
Keywords: Autism spectrum disorder; Bone density; Oxytocin; Peri-pubertal children
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: All subjects and all study staff except the pharmacist will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1. Intranasal Oxytocin (Experimental): Intranasal oxytocin spray (30 IU twice daily) for 12 months in the double-blinded phase followed by intranasal oxytocin spray (30 IU twice daily) for 6-months in the open-label phase
  Interventions: Drug: 1. Intranasal oxytocin spray; Drug: 3. Intranasal Oxytocin spray
- 2. Placebo (Placebo Comparator): Intranasal placebo spray (30 IU twice daily (total 60 IU per day) for 12 months followed by intranasal oxytocin spray (30 IU twice daily) for 6-months in the open-label phase
  Interventions: Drug: 2. Intranasal placebo spray; Drug: 3. Intranasal Oxytocin spray

INTERVENTIONS:
Drug: 1. Intranasal oxytocin spray — 30 IU, twice daily for 12 months in the experimental arm in double-blinded phase
  Arms: 1. Intranasal Oxytocin
Drug: 2. Intranasal placebo spray — 30 IU, twice daily for 12 months in the placebo comparator arm in double-blinded phase
  Arms: 2. Placebo
Drug: 3. Intranasal Oxytocin spray — 30 IU, twice daily for 6 months in both experimental and placebo comparator arm in open-label phase

SUMMARY:
This is a randomized, double blind, placebo-controlled study of the effects of intranasal oxytocin on bone health in children with autism spectrum disorder, ages 6-18 years old. Subjects will be randomized to receive intranasal oxytocin or placebo (30 IU, 2 times daily) for 12 months in the double-blind phase, followed by a 6-month open label phase during which all study subjects will receive intranasal oxytocin (30 IU, 2 times daily). Study visits include screening to determine eligibility, followed by study visits at baseline, week 2, and months 6, 12, 18 and phone calls every two weeks for the first two months and monthly thereafter for the duration of the study. Study assessments include history and physical examinations, anthropometric measurements, electrocardiogram (EKG), adverse event monitoring, laboratory tests for chemistries, hormones and biomarkers for bone metabolism, questionnaires regarding diet and exercise, and imaging to assess body composition, bone density and structure.

DETAILED DESCRIPTION:
The prevalence of autism spectrum disorder (ASD), a group of behaviorally-defined disorders characterized by impaired social interactions and verbal and non-verbal communication, is increasing among children. Studies have shown that children with ASD are at a higher risk for low bone mineral density and fractures. ASD is also characterized by low levels of oxytocin (OXT), a peptide hormone with prosocial effects. In addition, OXT promotes bone formation over resorption and low levels of OXT are associated with poor bone health. Hence, OXT administration represents a potential strategy for improving bone health in children with ASD, particularly during the childhood and adolescent years when bone accrual peaks.

The investigators aim to examine (i) whether intranasal OXT administration vs. placebo increases areal bone mineral density (BMD) and improves overall bone health in children with ASD, and (ii) other pathways whereby OXT may impact bone health favorably.

The investigators will enroll 96 participants 6-18 years old with ASD and randomize them into the intranasal oxytocin vs. placebo groups. The study subjects will undergo history and physical examinations, anthropometric measurements, electrocardiogram (EKG), adverse event monitoring, laboratory tests for chemistries, hormones and biomarkers for bone metabolism, questionnaires regarding diet and exercise, and imaging to assess body composition, bone density and structure.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 6 to 18 years old at Randomization
2. BMI greater than or equal to the 5th percentile
3. Expert clinical diagnosis of ASD
4. Availability of parent/guardian to provide informed consent

Exclusion Criteria:

1. Fragile X, tuberous sclerosis, and other single gene defects that are syndromic
2. Other conditions that may contribute to low bone density (e.g., hypogonadism)
3. Medications that may impact bone other than calcium or vitamin D supplementation, other than calcium or vitamin D supplementation, such as specific anti-seizure medications (Phenytoin, Phenobarbital), oral glucocorticoids, hormonal contraceptive injection (Medroxyprogesterone acetate (Depo-Provera)
4. Hyponatremia
5. Liver enzymes (AST, ALT, and Bilirubin) more than three times the upper limit of the normal range
6. Estimated glomerular filtration rate (eGFR) less than 60
7. Substance use disorder within the last 6 months
8. History of known coronary artery disease, heart failure, reduced ejection fraction, hypertrophic cardiomyopathy, ventricular arrhythmias, or prolonged QT (QTc greater than or equal to 480 msec)
9. Active seizures within 6 months preceding the Screening visit or the Baseline visit
10. Subjects who are pregnant, lactating, or who refuse contraception if sexually active
11. Subjects who have had previous treatment with OXT (within 2 months of Randomization)
12. Subjects who are not able to cooperate with medication administration, blood drawing, or imaging procedures despite behavior training
13. Caregivers who are unable to speak English, be consistently present at study visits to report on symptoms or, per the judgement of the data collection team, are unable to comply with the protocol
14. Any significant illness, condition, medication, or medical device that the Investigator determines could interfere with study participation and impact data collection or subject safety

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Difference between IN OXT vs placebo in 12-month change in whole body less head BMD Z-scores. | 12 months

SECONDARY OUTCOMES:
Difference between IN OXT vs placebo in 12-month change in areal BMD Z-score at the femoral neck. | 12 months
Difference between IN OXT vs placebo in 12-month change in radial and tibial cortical area and radial trabecular thickness. | 12 months
Difference between IN OXT vs placebo in 12-month change in radial and tibial failure load. | 12 months
Difference between IN OXT vs placebo in 12-month change in bone turnover markers, cortisol. | 12 months
Difference between IN OXT vs placebo in 12-month change in lean mass and muscle area | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Lawson, MD, Principal Investigator — Neuroendocrine Unit Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Virginia Medical Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No